CLINICAL TRIAL: NCT04477356
Title: The Effectiveness of Swim-up Versus Gradient Density for Sperm Preparation in Patients Undergoing Intrauterine Insemination: A Randomized Controlled Trial.
Brief Title: SU Versus GD for Sperm Preparation in IUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: Mỹ Đức Phú Nhuận Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS/BVMDPN/20/02
Record Dates: First submitted 2020-07-06; First posted 2020-07-20 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2022-12

CONDITIONS: Infertility
Keywords: Swim-up (SU); Gradient density (GD); IUI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The prepared sperms will be proceeded to medical doctor who will carry the IUI and have no information about the semen preparation step.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swim-up technique (SU) (Active Comparator): The SU method's principle is that the normal and highly motile sperm will move against the gravity and separate from the dead or abnormal sperms to swim up to the upper media culture layer.
  Interventions: Procedure: SU
- Density gradient centrifugation technique (DG) (Active Comparator): The DG method is based on the density in which mature and normal sperms are capable of passing through filtration layer to be isolated from dead or abnormal sperms in semen.
  Interventions: Procedure: DG

INTERVENTIONS:
Procedure: SU — Aliquot 1.2 ml Ferticult Flushing media (Fertipro, Belgium) into 14 ml tube and then gently add 1 ml semen sample to the bottom of the tube (in case of larger semen volume, use multiple 14 ml tubes). The tubes then will be hold at an angle of 45 degrees for 45-60 minutes at 37C. Collect 1 ml of supernatant and then wash with 2 ml Ferticult Flushing media by centrifugation at 1200 RPM for 10 minutes. Keeping 0.3 ml washed semen for IUI, sperm density counting. Prepared sperms will be transferred into uterus by soft catheter (Gynétics, Belgium).
  Arms: Swim-up technique (SU)
Procedure: DG — Add 1.5 ml Sil-select 90% first and then 1.5 ml Sil-select 45% (Fertipro, Belgium) into centrifuge tube, then gently add 1 - 1.5 ml semen on the top of Sil-select layer and centrifuge at 1200 RPM for 15 minutes. Discard upper layer, collect 0.5 ml lower layer into new tube and then wash with 2 ml Ferticult Flushing media at 1200 RPM for 10 minutes. Discard upper layer then collect 0.3 ml lower layer for IUI, sperm density counting. Prepared sperms will be transferred into uterus by soft catheter (Gynétics, Belgium).
  Arms: Density gradient centrifugation technique (DG)

SUMMARY:
Intrauterine insemination (IUI) is the first-line treatment for couples with unexplained and mild male factor infertility. The result of IUI depends on many factors including the sperm preparation techniques. Swim-up (SU) and Density Gradient (DG) are the two most commonly used techniques in sperm preparation for IUI. There is discussion about the effectiveness of these two techniques for IUI outcomes. The effectiveness of SU and DG methods on IUI success rate is not clearly understood and is controversial. This multicenter, randomized controlled trial will be conducted to determine which method (DG or SU) is better for IUI treatment.

DETAILED DESCRIPTION:
Potentially eligible patients will be given information about the study on day 2 or day 3 of the menstrual cycle, when the ovarian stimulation starts. Screening for eligibility will be performed by treating physicians on the day of IUI, after having obtained the semen qualified for inclusion criteria from the husband. Eligible participants will be invited to a full discussion with investigators about the study and will be given the informed consent form. Couples will have enough time to decide if they agree to participate in the study or not. Written informed consent will be obtained by the investigators from all couples prior to enrolment. When a participant signs an informed consent, she is considered to be enrolled in the study.

Eligible patients who have provided informed consent will be randomized in a 1:1 ratio to either SU or GD. Assignment to treatment allocation will be done via a web portal hosted by HOPE Research Center, Vietnam. The randomization schedule will be computer-generated at HOPE Research Center, with a permuted random block size of 2, 4, and 6. Blinding will not be possible due to the nature of interventions.

Ovarian stimulation will be performed by using human menopausal gonadotrophins (hMG) (IVF-M, LG Life science, Korea) and follicular development will be monitored by transvaginal ultrasound every 3 - 5 days begin on day 2 or day 3 of the menstrual cycle. An injection of human chorionic gonadotropin (hCG) (IVF-C 5000 IU, LG Life Science, Korea) will be given to trigger ovulation when the mean diameter of the dominant follicle reached ≥ 18 mm. Those who have more than 7 follicles ≥ 14 mm will be subjected to cancel or convert to IVM. IUI will be scheduled 36 - 38 hours after hCG injection.

A sperm sample will be obtained in the clinic by masturbation after 2-5 day of abstinence. Spoken and written instructions about the collection of the semen sample will be given in advance. The time between semen production and processing will be up to 1 hour. Sperm preparation will be performed after the patient agrees to participate in the study.

In couples allocated to the sperm swim-up technique (SU): the normal and highly motile sperm will move against the gravity and separate from the dead or abnormal sperms to swim up to the upper media culture layer In couples allocated to the sperm density gradient centrifugation technique (GD): the density in which mature and normal sperms are capable of passing through filtration layer to be isolated from dead or abnormal sperms in semen Prepared sperms will be transferred into uterus by soft catheter (Gynétics, Belgium). Luteal-phase support will be done with vaginal progesterone 400 mg per day (Cyclogest 200 mg, Actavis, UK) until 7th week of gestation. In both groups, clinicians who perform insemination will be blinded to the intervention.

The prepared sperms will be proceeded to medical doctor who will carry the IUI and have no information about the semen preparation step. After insemination, the patient will be asked to immobilize for 15 minutes. The patient will receive luteal phase support using vaginal micronized progesterone for 14 days. In both groups, blood hCG will be measured at day 14 after insemination, and positive results indicate biochemical pregnancy. If the gestational sac is observed with ultrasonography at week 7 after transferring, clinical pregnancy will be confirmed. At the 11th and 12nd weeks of gestation, participants will be referred to the Outpatient clinic, OB/GYN Department at My Duc hospital or at My Duc Phu Nhuan hospital for prenatal care until delivery. When the participant attends for delivery, data on labor and delivery, any complications experienced by participant, and the neonates will be collected. For those who cannot participate the prenatal care program at either the two hospitals, for any reasons, we will contact the participants via telephone/email monthly until delivery to collect data. We also ask these participants to scan their profile in every contact.

All analyses will be conducted on an intention-to-treat basis using the R statistical program The rate of live birth and the associated 95% confidence interval (CI) will be estimated and compared between groups using the exact method for binomial proportion.

Differences between groups in secondary outcome variables will be analyzed using Student t-test or Wilcoxon signed-rank test for normally distributed or skewed variables, and Fisher's exact test for categorical variables, and reported as relative risk (RR) with 95% CI. Besides that, we will conduct the subgroup analysis to compare the effectiveness of DG and that of SU for each of criteria within the following categories including causes of infertility, quality of pre-washing semen, and total number of post-washing motile sperms. For the number of motile sperms after washing, we divide it into 5 subgroups including < 1 million sperms, 1-5 million sperms, 5-10 million sperms, 10-20 million sperms, and > 20 million sperms.

For missing population characteristics, first, we will analyze by removing the missing data; then we perform multiple imputations of lost values and perform another analysis to estimate the certainty of these obtained results. In case of losing track of patients or making protocol mistakes, we will try performing sensitivity analysis to evaluate the effects of these factors in the study. A statistical analysis plan will be made and signed before data-lock.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IUI
* Undergone ≤ 2 previous IUI cycles
* Progressive motility (PR) before sperm preparation: ≥ 32%
* Sperm concentration before sperm preparation: ≥ 5 million/ml
* Total progressive motility sperm count before sperm preparation: > 5million
* Agree to participate in the study

Exclusion Criteria:

* Using frozen semen
* High viscosity semen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate | At 24 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 24 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. In the analysis for the primary endpoint, twin delivery will be considered.

SECONDARY OUTCOMES:
Total motile sperm count after sperm preparation | At 5 minutes after sperm preparation for IUI
  Total motile sperm count after sperm preparation, measured by million sperm
Biochemical pregnancy rate | At 14 days after insemination
  Biochemical pregnancy defined as a serum beta-hCG level greater than 25 mIU/ml at day 14 after insemination.
Clinical pregnancy rate | At 7 weeks of gestation
  Clinical pregnancy defined as the presence of at least one gestational sac on ultrasound at week 7 of gestation with the detection of heart beat activity, after insemination.
Ongoing pregnancy rate (OPR) | At the 12 weeks of gestation
  Ongoing pregnancy is defined as a living intrauterine fetus at the 12th week of gestation.
Ectopic pregnancy rate | At 5-7 weeks of gestation
  Ectopic pregnancy defined as a pregnancy in which implantation takes place outside the uterine cavity
Multiple pregnancy rate | At 7 weeks of gestation
  Multiple pregnancy defined as two or more gestational sacs or two or more positive heart beats by transvaginal sonography
Vanishing twin rate | In the first trimester pregnancy
  Vanishing twin defined as the spontaneous reduction of a fetus while still in uterus.
Miscarriage rate | Before 22 weeks of gestational age
  Miscarriage defined as spontaneous loss of a clinical pregnancy before week 22 of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.
Gestational age at delivery | At birth
  Gestational age at delivery.
Stillbirth rate | After 28 completed weeks of gestational age
  Stillbirth defined as the death of a fetus prior to the complete expulsion or extraction from its mother.
Preterm labor rate | At birth
  Preterm delivery is defined as any delivery at <24, <28, <32, <37 completed weeks' gestation
Spontaneous preterm birth rate | At birth
  Spontaneous preterm birth is defined as delivery spontaneously at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth rate | At birth
  Iatrogenic preterm birth is defined as delivery non-spontaneously at <24, <28, <32, <37 completed weeks
Birth weight | At birth
  Weight of newborn
Low birth weight rate | At birth
  Low birth weight is defined as <2500 gm
Very low birth weight rate | At birth
  Very low birth weight is defined as <1500 gm
High birth weight rate | At birth
  High birth weight is defined as >4000 gm
Very high birth weight rate | At birth
  Very high birth weight is defined as >4500 gm
1-minute Apgar score | 1 minute after delivery
  1-minute Apgar score (0-10 score)
5-minutes Apgar score | 5 minutes after delivery
  5-minutes Apgar score (0-10 score)
Admission to NICU rate | 7 days after delivery
  The admittance of the newborn to NICU
Congenital abnormalities rate | At birth
  Any congenital abnormalities detected in the newborn

CONTACTS AND LOCATIONS:
Locations (1):
- Dang Q Vinh, Hochiminh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duong TND, Dang VQ, Le TK, Vu ATL, Nguyen DL, Pham TD, Nguyen MT, Nguyen PTM, Vo TM, Nguyen CTH, Le PTB, Le AH, Tran CT, Mol BW, Vuong LN, Ho TM. Swim-up versus density gradients for sperm preparation in infertile couples undergoing intrauterine insemination: a randomized clinical trial. Hum Reprod. 2025 May 1;40(5):788-795. doi: 10.1093/humrep/deaf047. PMID 40135621